CLINICAL TRIAL: NCT03885401
Title: Enhanced Care Planning and Clinical-Community Linkages to Comprehensively Address the Basic Needs of Patients With Multiple Chronic Conditions
Brief Title: Enhanced Care Planning for Patients With Multiple Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HM20015553; 1R01HS026223-01A1 (AHRQ)
Record Dates: First submitted 2019-03-09; First posted 2019-03-21 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Multiple Chronic Conditions; Health Behavior; Mental Health; Social Determinants of Health
MeSH Terms: conditions — Multiple Chronic Conditions; Health Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is a clinician level randomized controlled trial. Sixty clinicians will be randomized to intervention (enhanced care planning for health behaviors, mental health, and social needs) or control condition (usual care). The investigators will randomly survey all patients with MCC from each clinicians' patient panel. Patients with at least one uncontrolled MCC will be randomly selected for inclusion until 10 patients are recruited from each clinician. The investigators will use hybrid implementation-effectiveness design to measure outcomes. Implementation outcomes include enhanced care plan completion; the prevalence of health behavior, mental health, and social needs; goals patients prioritize and how they want to address them; and the type, intensity, and follow-up of care team support provided to address patient goals. Effectiveness outcomes include the number of uncontrolled chronic conditions and patient reported physical, mental, and social health..
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind clinicians, patients, or patient navigators. Outcomes assessors (e.g. chart abstractors, database managers, and the researchers) will be blinded to condition when abstracting, entering, or assessing data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced care planning (Experimental): The intervention consists of two components - enhanced care planning and clinical-community linkages. The enhanced care plan is created using MOHR (https://myownhealthreport.org). MOHR screens patients for unhealthy behaviors, mental health needs, and social needs. Patients identify the needs they would like to address and create a care plan, which they update quarterly. A clinical navigator and community health worker (CHW) help patients address their care plans using clinical-community linkages, which has four components. First, clinicians and clinical navigators have a resource registry identifying community programs and support - No Wrong Door (NWD) and https://navigator.aafp.org/. Second, MOHR shares information (care plans, patient narrative, and patient progress) across clinical and community team members. Third, MOHR supports messaging and video visits for team members and patients. Finally, MOHR sends care team members quarterly patient progress updates.
  Interventions: Behavioral: Enhanced care planning
- Usual medical care (No Intervention): Clinicians randomized to the control condition will continue to provide "usual care." This includes current non-systematic assessment of health behaviors, mental health needs, and social needs. Neither clinicians nor patients will be eligible to receive CHW support or have access to NWD. Clinicians may refer some control patients to community programs as part of their current usual care. Control clinicians will be blinded as to which patients are included in the study. At the end of the study, the investigators will share with control clinicians our lessons learned, access to MOHR, and lists of useful community resources.

INTERVENTIONS:
Behavioral: Enhanced care planning — The intervention includes (1) screening for unhealthy behaviors, mental health needs, and social needs, (2) creation of a care plan, (3) quarterly updates to the plan, (4) a clinical navigator and community health worker to support accomplishing the care plan, (5) registry of community resources and programs, and (6) messaging and video-visit system for team members.
  Arms: Enhanced care planning

SUMMARY:
Patients with multiple chronic conditions (MCC) have a range of needs that extend beyond traditional medical care, including behavioral, mental health, and social needs. While primary care does its best to address these needs, few practices can undertake a systematic approach without broader health system and coordinated community support. Fortunately, communities and health systems are investing in new models of care to address these needs. New tools are emerging that allow for enhanced care planning to identify and prioritize patients' needs based on their values, preferences, social, and clinical context. Additionally, support systems to promote partnerships between patients and clinical and community care teams are emerging. Building on work occurring as part of the Richmond Accountable Health Community, the investigators propose to (a) evaluate the implementation of an enhanced care planning approach, paired with community-clinical linkages support to address health behavior, mental health, and social needs; (b) determine within a randomized controlled trial the benefit of this approach compared to usual care; and (c) assess which person, family, community, and system contextual factors that influence MCC.

DETAILED DESCRIPTION:
The number of patients in the United States with multiple chronic conditions (MCC) is growing. Many patients with poorly controlled MCC also have unhealthy behaviors, mental health challenges, and unmet social needs. Medical management of MCC may have limited benefit if patients are struggling to address these basic life needs. Health systems and communities increasingly recognize the need to address these issues and are experimenting with and investing in new models for connecting patients with needed services. Yet primary care clinicians, whose regular contact with patients makes them more familiar with patients' needs, are often not included in these systems. Responding to the Special Emphasis Notice NOT-HS-16-013, Optimizing Care for People Living with MCC through the Development of Enhanced Care Planning, the investigators propose a clinician-level randomized controlled trial to study how primary care clinicians can participate in these community and hospital solutions and whether doing so is effective in controlling MCC. This study will build on the Centers for Medicare and Medicaid Services (CMS)-funded Accountable Health Community (AHC) in Richmond, Virginia. Sixty clinicians in the Virginia Ambulatory Care Outcomes Research Network (ACORN) will be matched by age and sex and randomized to usual care (control condition) or enhanced care planning with clinical-community linkage support (intervention). From the electronic health record (EHR), clinicians will identify all patients with MCC, including cardiovascular disease or risks, diabetes, obesity, or depression. A baseline assessment will be mailed to 50 randomly selected patients; 10 respondents per clinician (600 patients total) with uncontrolled MCC will be randomly selected, with over-sampling of minorities. The intervention includes two components. First, an enhanced care planning tool called My Own Health Report (MOHR) will screen patients for health behavior, mental health, and social needs. Clinical navigator support will help patients prioritize needs, create care plans based on preferences, and write a personal narrative to guide the care team. Patients will update care plans quarterly. Second, community-clinical linkage support will include community resource registries, personnel to span settings (clinical navigators, community health workers), and care team coordination tools (sharing MOHR content, secure messaging, and virtual visits). The investigators will compare patient-level intervention and control outcomes to assess improvements in MCC outcomes (primary outcome) and self-reported PROMIS-29 measures (physical health, mental health, social wellbeing) six months and two years post-enrollment. the investigators will also conduct a mixed-methods, multilevel assessment of person-, family-, community-, and system-level contextual influences on implementation and effectiveness. Data sources will include EHR and MOHR data, chart reviews, patient surveys, field notes, and semi-structured interviews of patients, clinicians, and community stakeholders. If effective, this study will help inform efforts by primary care clinicians to participate in the growing number of AHC-like systems as a strategy to better control MCC.

ELIGIBILITY:
Inclusion Criteria:

* Two or more chronic conditions
* At least one uncontrolled condition
* Completes baseline survey

Exclusion Criteria:

* Participating in Richmond Accountable Health Community study
* Clinician excludes patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Enhanced care plan creation (implementation outcome) | Within 6 months of enrollment
  This outcome reports the percent of intervention patients who complete the creation of an enhanced care plan (numerator = intervention patients who create an enhanced care plan / denominator = all enrolled intervention patients).
Health behavior, mental health, and social needs | Within 6 months of enrollment
  This outcome will measure the number of health behavior, mental health, and social needs that patients have who complete an enhanced care plan. This is a frequency count of each specific need based on the health risk assessment output.
Referral to and connection to community resources (implementation outcome) | Over 2 years after enrollment
  This outcome will measure which community resources intervention patients are referred to for assistance with addressing health behaviors, mental health, and social needs. This is a frequency count of the number of intervention patients referred to each potential community resource.
Effectiveness - chronic condition control | 6 months after creating a care plan
  Percent of patients with an uncontrolled chronic condition for intervention patients versus usual care
Maintenance - chronic condition control | 2 years after creating a care plan
  Percent of patients with an uncontrolled chronic condition for intervention patients versus usual care
Effectiveness - quality of life: Patient Reported Outcomes Measurement Information System (PROMIS-29) | 6 months after creating a care plan
  Pre-post change in eight Patient Reported Outcomes Measurement Information System (PROMIS-29) domains for intervention patients versus usual care. Norm-based scores will be calculated for each domain on the PROMIS measures, so that a score of 50 represents the mean or average of the reference population. A score of 60 means that the person is one standard deviation above the reference population. Higher scores means that the patient is reporting greater symptoms. Scores will be calculated using the Healthmeasures Scoring Service (http://www.healthmeasures.net/score-and-interpret/calculate-scores).
Maintenance - quality of life: eight PROMIS-29 domains | 2 years after creating a care plan
  Pre-post change in eight PROMIS-29 domains for intervention patients versus usual care

CONTACTS AND LOCATIONS:
Overall Officials: Alex H Krist, MD MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krist AH, O'Loughlin K, Woolf SH, Sabo RT, Hinesley J, Kuzel AJ, Rybarczyk BD, Kashiri PL, Brooks EM, Glasgow RE, Huebschmann AG, Liaw WR. Enhanced care planning and clinical-community linkages versus usual care to address basic needs of patients with multiple chronic conditions: a clinician-level randomized controlled trial. Trials. 2020 Jun 11;21(1):517. doi: 10.1186/s13063-020-04463-3. PMID 32527322

DOCUMENTS (1):
  • Informed Consent Form (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT03885401/ICF_000.pdf